The value of end tidal capnograpy in the evaluation of mortality and morbidity in Patients who apply to the emergency department with complaints of gastrointestinal bleeding

## Statistical analysis

The obtained data were transferred to the SPSS 23.0 package program. Among the demographic data of the patients, categorical variables such as gender were calculated as number and percentage, and other numerical variables were calculated as mean and standard deviation. The evaluation of categorical variables in dependent groups was performed with McNemar test. In comparisons of continuous variables in dependent groups, conformity to normal distribution was evaluated by histogram curves and Shapiro-Wilks test. Paired t-test for dependent groups was used when the normal distribution condition was met, and Wilcoxon test was used when it was not met.

In all tests, p<0.05 was considered statistically significant.